CLINICAL TRIAL: NCT01813422
Title: A Double-blind, Randomized, Multi-center, Placebo-controlled, Parallel-group Study to Determine the Effects of Evolocumab (AMG 145) Treatment on Atherosclerotic Disease Burden as Measured by Intravascular Ultrasound in Subjects Undergoing Coronary Catheterization
Brief Title: GLobal Assessment of Plaque reGression With a PCSK9 antibOdy as Measured by intraVascular Ultrasound
Acronym: GLAGOV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120153; 2012-004208-37 (EudraCT Number)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; High Cholesterol; Elevated Cholesterol; Raised Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo to evolocumab administered by subcutaneous injection once a month for 76 weeks.
  Interventions: Drug: Placebo
- Evolocumab (Experimental): Participants received 420 mg evolocumab administered by subcutaneous injection once a month for 76 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha®
  Arms: Evolocumab
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
This study will evaluate whether low-density lipoprotein (LDL-C) lowering with evolocumab (AMG 145) results in greater change from baseline in percent atheroma volume (PAV) at week 78 than placebo in adults with coronary artery disease taking lipid lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for coronary angiography
* Subjects already taking statin therapy, niacin or ezetimibe at screening must have been on a stable dose for at least 4 weeks prior to screening LDL-C. Subjects not taking lipid-regulating therapy must enter the study via a lipid stabilization period. Subjects who are intolerant to statins must meet statin intolerance entry criteria
* Fasting LDL-C ≥ 80 mg/dL (2.07 mmol/L) with or without additional risk factors, or, LDL-C ≥ 60 -< 80 mg/dL (1.55-2.07 mmol/L) in the presence of one major or three minor risk factors

Subjects must meet the following criteria at the qualifying coronary catheterization procedure:

* Evidence of coronary heart disease (at least one lesion in a native coronary artery that has > 20% reduction in lumen diameter) or prior percutaneous intervention (PCI)
* Left main coronary artery < 50% reduction in lumen diameter by visual estimation
* Target coronary artery for IVUS must be accessible to the IVUS catheter, must not have a > 50% reduction in lumen diameter within the target segment (and at least 40 mm in length); cannot have undergone prior PCI or coronary artery bypass graft (CABG) and is not a candidate for intervention over the next 18 months. It may not be a bypass graft, bypassed vessel or culprit vessel for previous myocardial infarction (MI).

Exclusion Criteria:

* Coronary artery bypass graft surgery < 6 weeks prior to the qualifying IVUS
* New York Heart Association (NYHA) III or IV heart failure, or last known left ventricular ejection fraction less than 30%
* Uncontrolled cardiac arrhythmia that is not controlled by medications in the 3 months prior to randomization
* Known hemorrhagic stroke
* Uncontrolled hypertension at randomization
* Fasting Triglycerides ≥ 400 mg/dL (4.5 mmol/L) at screening
* Type 1 diabetes or poorly controlled type 2 diabetes (hemoglobin A1c [HbA1c] > 9%) at screening.
* Moderate to severe renal dysfunction (estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73m²) at screening.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (200):
- United States (57):
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Torrance, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hammond, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bay City, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Marquette, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Ridgewood, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Hillsboro, Oregon
  - Research Site, Springfield, Oregon
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
- Argentina (7):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
- Australia (13):
  - Research Site, Concord, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Bedford Park, South Australia
  - Research Site, Epping, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Nedlands, Western Australia
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Lodelinsart
- Brazil (6):
  - Research Site, Cariacica, Espírito Santo
  - Research Site, Goiânia, Goiás
  - Research Site, Curitiba, Paraná
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, São Paulo
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (2):
  - Research Site, Temuco, Cautín
  - Research Site, Santiago
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
- Denmark (2):
  - Research Site, Aarhus N
  - Research Site, Odense C
- France (6):
  - Research Site, Besançon
  - Research Site, Chambray-lès-Tours
  - Research Site, Créteil
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pessac
- Germany (6):
  - Research Site, Aachen
  - Research Site, Essen
  - Research Site, München
  - Research Site, Neuss
  - Research Site, Regensburg
  - Research Site, Ulm
- Greece (3):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
- Research Site, Reykjavik, Iceland
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Israel (3):
  - Research Site, Hadera
  - Research Site, Jerusalem
  - Research Site, Rehovot
- Italy (5):
  - Research Site, Novara
  - Research Site, Roma
  - Research Site, Rozzano MI
  - Research Site, Sesto San Giovanni (MI)
  - Research Site, Torino
- Malaysia (2):
  - Research Site, Kuantan, Pahang
  - Research Site, George Town
- Mexico (6):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Querétaro City, Querétaro
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Culiacán, Sinaloa
  - Research Site, Aguascalientes
  - Research Site, Puebla City
- Netherlands (11):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Leeuwarden
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Venlo
  - Research Site, Zwolle
- Norway (2):
  - Research Site, Oslo
  - Research Site, Tromsø
- Philippines (2):
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (5):
  - Research Site, Chrzanów
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Kemerovo
  - Research Site, Moscow
- Research Site, Singapore, Singapore
- South Africa (6):
  - Research Site, Boksburg, Gauteng
  - Research Site, Centurion, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Kuils River, Western Cape
  - Research Site, Pinelands, Cape Town, Western Cape
  - Research Site, Somerset West, Western Cape
- South Korea (3):
  - Research Site, Daejeon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Málaga, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Madrid
- Sweden (6):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Lund
  - Research Site, Örebro
  - Research Site, Solna
  - Research Site, Stockholm
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Sankt Gallen
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
- Research Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJ, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Scott R, Ungi I, Podolec J, Ophuis AO, Cornel JH, Borgman M, Brennan DM, Nissen SE. Effect of Evolocumab on Progression of Coronary Disease in Statin-Treated Patients: The GLAGOV Randomized Clinical Trial. JAMA. 2016 Dec 13;316(22):2373-2384. doi: 10.1001/jama.2016.16951. PMID 27846344
- [Background] Nicholls SJ, Puri R, Anderson T, Ballantyne CM, Cho L, Kastelein JJP, Koenig W, Somaratne R, Kassahun H, Yang J, Wasserman SM, Honda S, Shishikura D, Scherer DJ, Borgman M, Brennan DM, Wolski K, Nissen SE. Effect of Evolocumab on Coronary Plaque Composition. J Am Coll Cardiol. 2018 Oct 23;72(17):2012-2021. doi: 10.1016/j.jacc.2018.06.078. PMID 30336824
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Puri R, Nissen SE, Somaratne R, Cho L, Kastelein JJ, Ballantyne CM, Koenig W, Anderson TJ, Yang J, Kassahun H, Wasserman SM, Scott R, Borgman M, Nicholls SJ. Impact of PCSK9 inhibition on coronary atheroma progression: Rationale and design of Global Assessment of Plaque Regression with a PCSK9 Antibody as Measured by Intravascular Ultrasound (GLAGOV). Am Heart J. 2016 Jun;176:83-92. doi: 10.1016/j.ahj.2016.01.019. Epub 2016 Feb 17. PMID 27264224
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 163 centers in 30 countries in Europe, North America, Asia Pacific, and Latin America. The first participant was enrolled on 18 April 2013 and the last participant enrolled on 12 January 2015.
Pre-assignment Details: Participants who met all entry criteria were randomized 1:1 to receive evolocumab 420 mg once monthly (QM) subcutaneous (SC) or placebo QM SC for 76 weeks. Randomization was stratified by region.
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 486 | 484
Received Treatment | 484 | 484
Completed | 466 | 468
Not Completed | 20 | 16
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Death | 2 | 3
Not completed — Sponsor Decision | 2 | 1
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 486 | 484 | 970
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.8) | 59.8 (9.6) | 59.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 135 | 270
  Male | 351 | 349 | 700
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 34 | 58
  Not Hispanic or Latino | 462 | 450 | 912
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 17 | 14 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 4 | 9
  White | 453 | 456 | 909
  Multiple | 6 | 7 | 13
  Other | 3 | 2 | 5
Stratification Factor: Geographical Region [Number; unit: participants]
  North America | 88 | 86 | 174
  Europe | 332 | 332 | 664
  Latin America | 16 | 15 | 31
  Asia Pacific | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Atheroma Volume at Week 78
Description: Intravascular ultrasound (IVUS) was used to visualize the extent of atherosclerotic plaques in the coronary artery lumen. The extent of atherosclerosis was expressed as percent atheroma volume (PAV) in a ≥ 40 mm segment of one targeted (imaged) coronary artery, calculated as the percentage of the total vessel volume occupied by atheroma.
Time Frame: Baseline and week 78
Population: Randomized participants who received at least 1 dose of study drug, with a baseline IVUS and an IVUS measurement conducted after week 52 (IVUS analysis set)
Measure: Least Squares Mean (Standard Error); unit: percent atheroma volume
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 423 | 423
percent atheroma volume | 0.053 (0.189) | -0.955 (0.190)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for the treatment group, the geographic region stratification factor, and baseline PAV; LS Mean Treatment Difference = -1.007, 95% CI 2-sided [-1.375 to -0.640], Standard Error of Mean 0.187 — Treatment difference uses placebo as the reference

2. Secondary Outcome: Change From Baseline in Total Atheroma Volume at Week 78
Description: Intravascular ultrasound (IVUS) was used to visualize the extent of atherosclerotic plaques in the coronary artery lumen. Total atheroma volume (TAV) in a ≥ 40 mm segment of the targeted coronary artery was calculated as the average plaque area over the number of images that were evaluated by IVUS multiplied by the median vessel length to compensate for differences in segment length between participants.
Time Frame: Baseline and week 78
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm³
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 423 | 423
mm³ | -0.910 (1.214) | -5.799 (1.216)
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for the treatment group, the geographic region stratification factor, and baseline TAV; LS Mean Treatment Difference = -4.889, 95% CI 2-sided [-7.247 to -2.531], Standard Error of Mean 1.201 — Treatment difference uses placebo as the reference

3. Secondary Outcome: Percentage of Participants With Regression in Percent Atheroma Volume
Description: Intravascular ultrasound (IVUS) was used to visualize the extent of atherosclerotic plaques in the coronary artery lumen. The extent of atherosclerosis was expressed as percent atheroma volume (PAV) in a ≥ 40 mm segment of one targeted (imaged) coronary artery, calculated as the percentage of the total vessel volume occupied by atheroma.
  Regression in PAV was defined as any reduction from baseline in PAV.
Time Frame: Baseline and week 78
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 423 | 423
percentage of participants | 47.3 [42.6 to 52.0] | 64.3 [59.6 to 68.7]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Based on CMH test stratified by geographic region; Treatment Difference = 17.0, 95% CI 2-sided [10.3 to 23.5] — Treatment difference uses placebo as the reference

4. Secondary Outcome: Percentage of Participants With Regression in Total Atheroma Volume
Description: Intravascular ultrasound (IVUS) was used to visualize the extent of atherosclerotic plaques in the coronary artery lumen. Total atheroma volume (TAV) in a ≥ 40 mm segment of the targeted coronary artery was calculated as the average plaque area over the number of images that were evaluated by IVUS multiplied by the median vessel length to compensate for differences in segment length between participants.
  Regression in TAV was defined as any reduction from baseline in TAV.
Time Frame: Baseline and week 78
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 423 | 423
percentage of participants | 48.9 [44.2 to 53.7] | 61.5 [56.7 to 66.0]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Based on CMH test stratified by geographic region; Treatment Difference = 12.5, 95% CI 2-sided [5.8 to 19.1] — Treatment difference uses placebo as the reference

ADVERSE EVENTS:
Time Frame: From first dose of study drug until week 80
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab
Serious Adverse Events (participants affected / at risk) | 142/484 | 135/484
Other Adverse Events (participants affected / at risk) | 120/484 | 114/484
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=484) | Evolocumab (N=484)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 6
Angina pectoris (Cardiac disorders) | 11 | 17
Angina unstable (Cardiac disorders) | 7 | 8
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 5 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 6
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 13 | 7
Coronary artery dissection (Cardiac disorders) | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 3
Coronary artery stenosis (Cardiac disorders) | 5 | 3
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Palpitations (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinoatrial block (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 11
Oedema peripheral (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular stent restenosis (General disorders) | 2 | 3
Vascular stent stenosis (General disorders) | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Gallbladder enlargement (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Eye infection toxoplasmal (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyonephrosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Arteriogram coronary (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer stage I, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chemodectoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 1
Device leakage (Product Issues) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Mental status changes (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Cervical polyp (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Coronary revascularisation (Surgical and medical procedures) | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Mammoplasty (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 0 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Vasoconstriction (Vascular disorders) | 0 | 1
Vessel perforation (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=484) | Evolocumab (N=484)
Angina pectoris (Cardiac disorders) | 32 | 21
Chest pain (General disorders) | 26 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 34
Headache (Nervous system disorders) | 29 | 19
Hypertension (Vascular disorders) | 34 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.